CLINICAL TRIAL: NCT05711446
Title: A Randomized Trial of Double Voiding Versus Usual Voiding to Reduce the Incidence of Urinary Tract Infections in Kidney Transplant Recipients
Brief Title: Double Voiding and Post-transplant UTI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-03024620
Record Dates: First submitted 2022-12-20; First posted 2023-02-03 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Urinary Tract Infections; Kidney Transplant; Complications
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double Voiding (Experimental): The participant will be instructed to void twice.
  Interventions: Other: Double Voiding
- Regular Voiding (Active Comparator): The participant will be instructed to void normally.
  Interventions: Other: Regular Voiding

INTERVENTIONS:
Other: Double Voiding — Participant will be instructed to void twice.
  Arms: Double Voiding
Other: Regular Voiding — Participant will void as usual
  Arms: Regular Voiding

SUMMARY:
Urinary tract infections (UTI) are common in kidney transplant recipients and are an important cause of illness and hospital admissions. Past studies have shown that about 1 out of 5 of newly transplanted patients develop UTI within their first 3 months of transplantation. Such UTIs increase the risk for blood stream infection and acute rejection of the kidney, Improvements in urinary voiding techniques may reduce the frequency of UTI. The purpose of this study is to evaluate the benefits of "double voiding" in kidney transplant recipients.

DETAILED DESCRIPTION:
Urinary tract infections are common in kidney transplant recipients and are an important cause of morbidity and hospital readmissions. Several risk factors for UTI, both modifiable and unmodifiable, have been described in the literature. In normal (non-transplant) individuals, because of the anatomy of the ureter insertion into the bladder that creates a valve-like effect during voiding, reflux of urine into the kidney is prevented . However, after kidney transplantation, urine refluxing into the transplanted kidney is common. Depending on the surgical technique used for connecting the transplant ureter to the urinary bladder, reflux may occur in up to 79% of kidney transplant recipients. In addition, the routine usage of ureteral stents (double J stents) for the first 4-6 weeks after transplantation results in reflux. Vesicoureteral reflux increases the risk of UTI Double voiding, a process of passing urine more than once each time, is a technique that may assist the bladder to empty more effectively when urine is left in the bladder. By reducing the amount of left-over urine in the bladder after each void, double voiding may help reduce the incidence of UTI in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* All adult kidney transplant recipients who undergo routine follow-up at the New York Presbyterian - Weill Cornell Medicine (NYP-WCM) Transplant Clinic.

Exclusion Criteria:

* Kidney transplant recipients who are discharged after a transplant with an indwelling catheter (Foley)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of UTI's | First 3 months of transplantation
  UTI will be defined as a clean catch urine bacterial culture that is reported as anything other than "<1000 CFU/ml (Colony Forming Unit / Milliliter)- Negative". Clean catch urine cultures are done at each follow-up visit as a standard of care, irrespective of patient symptoms. Hence the outcome will include both asymptomatic and symptomatic UTIs.

SECONDARY OUTCOMES:
Time to first bacterial culture | First 3 months of transplantation
  Time will be measured in days
Number of UTI episodes | First 3 months of transplantation
Bacterial colony count of each positive urine culture | First 3 months of transplantation
Number of incidences of bacteremia | First 3 months of transplantation
Number of hospital admissions | First 3 months of transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Muthukumar Thangamani, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College / NY Presbyterian, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee JR, Bang H, Dadhania D, Hartono C, Aull MJ, Satlin M, August P, Suthanthiran M, Muthukumar T. Independent risk factors for urinary tract infection and for subsequent bacteremia or acute cellular rejection: a single-center report of 1166 kidney allograft recipients. Transplantation. 2013 Oct 27;96(8):732-8. doi: 10.1097/TP.0b013e3182a04997. PMID 23917724
- [Background] Sarier M, Yayar O, Yavuz A, Turgut H, Kukul E. Update on the Management of Urological Problems Following Kidney Transplantation. Urol Int. 2021;105(7-8):541-547. doi: 10.1159/000512885. Epub 2021 Jan 28. PMID 33508852
- [Background] Garcia-Roig ML, Kirsch AJ. Urinary tract infection in the setting of vesicoureteral reflux. F1000Res. 2016 Jun 30;5:F1000 Faculty Rev-1552. doi: 10.12688/f1000research.8390.1. eCollection 2016. PMID 27408706
- [Background] Staessen J, Celis H, De Cort P, Fagard R, Thijs L, Amery A. Methods for describing the diurnal blood pressure curve. J Hypertens Suppl. 1991 Dec;9(8):S16-8. PMID 1795193